CLINICAL TRIAL: NCT05133622
Title: Muscle Strength, Muscle Endurance, Flexibility and Balance in Young Healthy Adults After COVID-19 Infection
Brief Title: Physical Fitness in Young Healthy Adults After COVID-19 Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Ozlem Yuruk, Assoc. Prof., Baskent University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KA21/233
Record Dates: First submitted 2021-11-23; First posted 2021-11-24 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
Keywords: COVID-19; Flexibility; Physical Fitness; Muscle strength; postural balance
MeSH Terms: conditions — COVID-19 | interventions — Pliability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Covid-19 group (Active Comparator): Individuals between the ages of 20-30 Individuals who were diagnosed with COVID-19 positive in the last 3-10 months and were treated with home isolation and whose last PCR test was negative Individuals who had not to get vaccinated Individuals whose physical activity level is between 600-3000 MET min/week according to "International Physical Activity Questionnaire-Short form (IPAQ-SF)" (sedentary)
  Interventions: Other: Physical Activity Level; Other: Evaluation of knee extension and elbow flexion muscle strength; Other: Evaluation of functional strength of trunk muscles; Other: Muscle Endurance; Other: Flexibility; Other: Balance; Other: Fatigue
- Control group (Active Comparator): Individuals between the ages of 20-30 Individuals who have not been diagnosed with COVID-19 positive Individuals who had not to get vaccinated Individuals whose physical activity level is between 600-3000 MET min/week according to the IPAQ-SF (sedentary)
  Interventions: Other: Physical Activity Level; Other: Evaluation of knee extension and elbow flexion muscle strength; Other: Evaluation of functional strength of trunk muscles; Other: Muscle Endurance; Other: Flexibility; Other: Balance; Other: Fatigue

INTERVENTIONS:
Other: Physical Activity Level — IPAQ-SF assesses the physical activity levels of the individuals. The short form of the questionnaire consists of seven questions and provides information about the time spent sitting, walking, moderately vigorous, and vigorous activities. In scoring, below 600 MET-min/week indicates individuals who are not physically active, 600-3000 MET-min/week values indicate low physical activity levels, and 3000 MET-min/week and above values indicate individuals with high physical activity levels. In our study, sedentary individuals who receive 600-3000 MET-min/week from the questionnaire will be included
Other: Evaluation of knee extension and elbow flexion muscle strength — To measure the knee extension strength, the individual brings the knee from 90 degrees flexion to full extension in sitting. To standardize the test, the lower extremities will be fixed of the chair with a belt, allowing full extension of the knee. Three measurements will be performed from the distal tibia with a dynamometer, and the score will be recorded in Newtons.
  Elbow flexion will also be measured in a sitting position in a chair. To standardize the given resistance, the upper extremity of the individual will be fixed to the arm support of the chair, allowing elbow flexion with a belt. During the measurement, the individual will try to flex the forearm in supination. Meanwhile, three measurements will be taken from the distal forearm with a dynamometer. The average score will be recorded in Newtons.
Other: Evaluation of functional strength of trunk muscles — Sit-ups test: The sit-ups test is a measure the endurance of the abdominal and hip-flexor muscles. The physiotherapist will fix the feet and ask the individuals to do trunk flexion in the knee flexion position. The number of movements performed for 30 seconds will be recorded.
  Push-ups test: The test will be in the prone position, with the hands at shoulder level and the elbows flexed, positioned near to the body. Individuals will raise the head, shoulders, and trunk from the ground with their elbows in full extension. The test is performed with the knees in full extension for men and modified knees in flexion for women. The number of movements performed for 30 seconds will be recorded.
Other: Muscle Endurance — Lateral bridge test: Lateral bridge test involves static, isometric contractions of the lateral muscles on each side of the trunk that stabilizes the spine.
  Modified Biering-Sorensen test: The test measuring how many seconds the individual can keep the unsupported upper body horizontal, while placed prone with the buttocks and legs fixed to the couch by three wide canvas straps and the arms folded across the chest.
  Trunk flexors endurance test: Trunk flexion test involving a static, isometric contraction of the anterior muscles, stabilizing the spine until the individual exhibits fatigue. The researcher stops the test when the individual cannot hold the assumed position.
  Prone bridge test: The prone bridge test measures the muscular endurance of the abdominal muscles.
Other: Flexibility — Back scratch test The back-scratch test evaluates upper extremity flexibility. The individual will externally rotate one arm over her/his shoulder to reach the lowest point on the back with the palm facing the back. The other extremity reaches the highest point on the back with the palm facing forward by internal rotation of the other arm. The distance between the middle fingers of both hands will be measured with a tape measure.
  Sit and reach test Sit and reach test evaluates lower extremity flexibility. In the test, a sit and reach board is used. The "0" reference point is taken as the 25 cm inner part where the feet are placed on the sit and reach the board. The part closer to the individual from the reference point shows negative values, and the part towards the far side shows positive values. Individuals will reach as far as with their fingertips by placing their feet on a sit-and-reach board.
Other: Balance — Single leg stance test Individuals bend one knee and place the sole on the other thigh and maintain their balance in this position. The test will be performed separately for the right and left extremities with eyes open and closed. The single-leg stance balance time was recorded as seconds (Linda,2013).
  Functional reach test The functional reach test evaluates dynamic balance and limit of stability. This test measures the distance between the length of an outstretched arm in a maximal forward reach from standing while maintaining a fixed base of support. The scoring record is centimeter. Higher scores indicate a good level of balance (Lin,2012).
Other: Fatigue — Individuals will score perceived fatigue during walking and running activities with the Modified Borg Scale. According to the scale, "0" indicates no fatigue, and a score of "10" indicates unbearable fatigue (Borg,1987).

SUMMARY:
Purpose:

The aim of this study is to evaluate muscle strength, muscle endurance, flexibility, and balance in individuals after mild COVID-19 infection and compare them with healthy individuals.

Methods:

A total of 118 individuals, 59 individuals between the ages of 18-30 who had COVID-19 (not vaccinated) and 59 individuals who did not, will be included in the study. Lower and upper extremity muscle strength, flexibility, and static and dynamic balances of the individuals will be evaluated and compared with the control group. The descriptive characteristics of the individuals will be recorded. The physical activity level of the individuals will be determined by the Short Form of International Physical Activity Questionnaire. The strength of knee extension and elbow flexion will be evaluated with a dynamometer, and functional trunk strength will be evaluated with sit-ups and push-ups tests. Lateral bridge test, modified Biering-Sorensen test, trunk flexors endurance test, and prone bridge test will be used to evaluate muscle endurance. Participants will perform sit and reach test and back scratch test for flexibility. The one-leg stance test and the functional reach test will be used to evaluate static and dynamic balance. The level of fatigue experienced by individuals during walking and running will score according to the Modified Borg Scale.

Results:

The SPSS for Windows 19.0 (IBM SPSS Statistics for Windows, Armonk, NY: IBM Corp.) will be used for data analysis. The data will be expressed as mean standard deviation (x±SD) and percentage (n%). The homogeneity of the groups will be evaluated with the Levene Test. Between groups, muscle strength, flexibility, and balance values will be compared using the "Mann Whitney-U" Test. The statistical significance level will be accepted as a p <0.05 value.

Conclusion:

The researchers will discuss the results in light of the recent literature.

DETAILED DESCRIPTION:
Introduction Pandemic is the general name given to epidemic diseases that spread and affect more than one country in the world. Most recently Coronavirus Disease 2019 (COVID-19) had a place among the epidemic diseases (Pollard, 2020). Although COVID-19 is involved in the primary respiratory system as acute respiratory distress syndrome, it also affects the cardiovascular and neurological systems (Guan,2020). The most common symptoms of COVID-19 infection are fever, cough, dyspnea, muscle pain, and fatigue. Infection can be seen in all age groups, especially in the elderly. The symptoms and course of the disease differ in children, young and older adults.

COVID-19 infection can be categorized clinically as mild, moderate, or severe (critical illness). The disease affects 80% of individuals with a mild/moderate clinical condition. Patients with mild symptoms and no pneumonia are in this group. Severe illness is seen with symptoms such as dyspnea, hypoxia, and affects more than 50% of the lungs in 24-48 hours. Approximately 14% of patients are in this group. Critical illness is seen at a rate of 2%. Patients should be followed in the intensive care unit because of a severe clinical picture such as respiratory failure, shock, and multi-organ failure (Mizumoto,2020).

Due to its effects on the pulmonary, cardiovascular and neurological systems, COVID-19 causes the physical functions of individuals to be adversely affected (Lau, 2005; Fiani, 2020). In the peripheral nervous system involvement, there are symptoms such as musculoskeletal pain, paresthesia, ataxia, and muscle weakness. In central nervous system involvement, there are findings such as headache and vertigo (Stevens, 2007).

When all these symptoms that occur with COVID-19 infection are combined with the negative effects of isolation and inactivity, it has been observed that physical fitness decreases in individuals (Pinho,2020).

In the literature, various studies evaluated physical fitness in middle-aged and elderly individuals who have had COVID-19 (Pinho,2020; Rooney 2020). These studies show that aerobic endurance and functional capacity of individuals decreased after COVID-19 infection (Rooney,2020). Some studies reported there is a decrease in muscle strength (Lee,2020; Carfi,2020).

Individuals may also experience decreased muscle strength, endurance, flexibility, and balance skills due to physical inactivity and disease (Pinho,2020; Rooney 2020). A decrease in muscle strength and endurance causes difficulty and fatigue in daily activities, decreased flexibility leads to musculoskeletal pain and predisposition to injuries, and impaired balance leads to loss of skills in daily living activities such as standing, walking, and climbing stairs (Pinho,2020; Biddle,2017). There were only a few studies show that isometric and concentric muscle strength and performance are negatively affected in individuals receiving acute care in the hospital (Carfi,2020; Vaes, 2020; Baririch,2021). Paneroni et al. reported that the quadriceps femoris muscle lost 86% and the biceps brachial muscle 73% of strength, in individuals aged 40-88 years in acute care (with moderate or severe COVID-19 infection). The authors compared the muscle strength and exercise tolerance with norm values and did not include a healthy control group. Baricich et al., examined the physical performance of 204 individuals with a mean age of 57.9 years, who were treated for COVID-19, were discharged 3-6 months ago. The authors observed that the balance, lower extremity strength, and walking capacity of individuals decreased.

As can be seen, the negative effects of COVID-19 infection on the pulmonary, cardiovascular, and neurological systems and the restriction of physical activity due to the pandemic process lead to a decrease in some physical fitness parameters (Franco, 2021). In the literature, some studies examined physical fitness parameters such as aerobic capacity and muscular strength in middle-aged or elderly patients receiving acute care in hospitals. These studies show that the aerobic capacity and muscular strength of individuals with severe exposure decrease. However, there are no studies on physical fitness parameters such as muscle strength, endurance, flexibility, and balance of young older adults who had mild disease. In addition, no comparison was made with a control group consisting of healthy individuals. This study aims to evaluate muscle strength, muscle endurance, flexibility, and balance in individuals with mild or moderate COVID-19 infection and compare them with healthy individuals.

MATERIALS AND METHODS Study Design The study will conduct on the Baskent University Faculty of Health Sciences Physiotherapy and Rehabilitation Department between December 2021 and February 2022. Ethics Committee of Baskent University Medicine and Health Sciences Research and Non-Interventional Clinical Research approved the study (project no: 21/93). Individuals participating in the study read and signed the informed consent form.

Participants

Individuals who are a student at Baskent University or working as health personnel at Baskent University Hospitals will be included in the study. There are two groups in the study:

Group 1: Individuals with COVID-19 infection and taking medication with home isolation Group 2: Healthy individuals without COVID-19 infection (Control group) The sample size was calculated with the G Power Version 3.1.9.5 (Universität Kiel, Kiel, Germany) program with 80% power and 0.05 margin of error, and it was found that a total of 118 individuals, 59 individuals in each group, should be included in the study.

Methods The individuals participating in the study will be evaluated with the pandemic rules at Baskent University Faculty of Health Sciences and Baskent Hospitals.

Socio-demographic Variable Descriptive and clinical characteristics of the individuals participating in the study such as age, gender, weight, height, occupation, and smoking status will be recorded.

Physical Activity Level IPAQ-SF assesses the physical activity levels of the individuals. The short form of the questionnaire consists of seven questions and provides information about the time spent sitting, walking, moderately vigorous, and vigorous activities. In scoring, below 600 MET-min/week indicates individuals who are not physically active, 600-3000 MET-min/week values indicate low physical activity levels, and 3000 MET-min/week and above values indicate individuals with high physical activity levels. In our study, sedentary individuals who receive 600-3000 MET-min/week from the questionnaire will be included (Craig,2003; Saglam,2010).

Evaluation of knee extension and elbow flexion muscle strength The strength of the quadriceps femoris and the biceps brachii will be evaluated bilaterally with a muscle strength dynamometer (Manual Muscle Tester 01165, Lafayette Instrument, USA). The literature was based on the selection of these muscles for evaluation (Paneroni,2021).

To measure the knee extension strength, the individual brings the knee from 90 degrees flexion to full extension in sitting. To standardize the test, the lower extremities will be fixed of the chair with a belt, allowing full extension of the knee. Three measurements will be performed from the distal tibia with a dynamometer, and the score will be recorded in Newtons.

Elbow flexion will also be measured in a sitting position in a chair. To standardize the given resistance, the upper extremity of the individual will be fixed to the arm support of the chair, allowing elbow flexion with a belt. During the measurement, the individual will try to flex the forearm in supination. Meanwhile, three measurements will be taken from the distal forearm with a dynamometer. The average score will be recorded in Newtons.

Evaluation of functional strength of trunk muscles Sit-ups test: The sit-ups test is a measure the endurance of the abdominal and hip-flexor muscles. The physiotherapist will fix the feet and ask the individuals to do trunk flexion in the knee flexion position. The number of movements performed for 30 seconds will be recorded.(Bliss, 2005, McGill, 2006).

Push-ups test: The test will be in the prone position, with the hands at shoulder level and the elbows flexed, positioned near to the body. Individuals will raise the head, shoulders, and trunk from the ground with their elbows in full extension. The test is performed with the knees in full extension for men and modified knees in flexion for women. The number of movements performed for 30 seconds will be recorded.

Muscle Endurance Static endurance of trunk muscles is evaluated according to McGill protocol (McGill,2006). In the measurements, the test score is recorded time recorded in seconds. The researcher stops the test when the individual deteriorates or does not continue.Higher scores indicate a good level of endurance.

Lateral bridge test: Lateral bridge test involves static, isometric contractions of the lateral muscles on each side of the trunk that stabilizes the spine.

Modified "Biering-Sorensen" test: The test measuring how many seconds the individual can keep the unsupported upper body (from the upper border of the iliac crest) horizontal, while placed prone with the buttocks and legs fixed to the couch by three wide canvas straps and the arms folded across the chest.

Trunk flexors endurance test: Trunk flexion test involving a static, isometric contraction of the anterior muscles, stabilizing the spine until the individual exhibits fatigue. The researcher stops the test when the individual cannot hold the assumed position.

Prone bridge test: The prone bridge test measures the muscular endurance of the abdominal muscles.

Flexibility Back scratch test The back-scratch test evaluates upper extremity flexibility. The individual will externally rotate one arm over her/his shoulder to reach the lowest point on the back with the palm facing the back. The other extremity reaches the highest point on the back with the palm facing forward by internal rotation of the other arm. The distance between the middle fingers of both hands will be measured with a tape measure. If the middle fingers do not touch each other, the distance between them is recorded as a minus value in centimeters, if fingers can reach completely, as a zero value, if the fingers cross each other, as a positive value in centimeters (Heyward, 2002).

Sit and reach test Sit and reach test evaluates lower extremity flexibility. In the test, a sit and reach board is used. The "0" reference point is taken as the 25 cm inner part where the feet are placed on the sit and reach the board. The part closer to the individual from the reference point shows negative values, and the part towards the far side shows positive values. Individuals will reach as far as with their fingertips by placing their feet on a sit-and-reach board. The test is repeated three times. The average score is recorded (Heyward, 2002).

Balance Single leg stance test Individuals bend one knee and place the sole on the other thigh and maintain their balance in this position. The test will be performed separately for the right and left extremities with eyes open and closed. The test score will recorded as seconds (Linda,2013).

Functional reach test The FRT evaluates dynamic balance and limit of stability. This test measures the distance between the length of an outstretched arm in a maximal forward reach from standing while maintaining a fixed base of support. The scoring record is centimeter (Lin,2012).

Fatigue Individuals will score perceived fatigue during walking and running activities with the Modified Borg Scale. According to the scale, "0" indicates no fatigue, and a score of "10" indicates unbearable fatigue (Borg,1987).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for individuals diagnosed with COVID-19 (Pinho,2020):

* Individuals between the ages of 20-30
* Individuals who were diagnosed with COVID-19 positive in the last 3-10 months and were treated with home isolation and whose last PCR test was negative
* Individuals who had not to get vaccinated
* Individuals whose physical activity level is between 600-3000 MET min/week according to "International Physical Activity Questionnaire-Short form (IPAQ-SF)" (sedentary)

Inclusion criteria of healthy individuals (Control group):

* Individuals between the ages of 20-30
* Individuals who have not been diagnosed with COVID-19 positive
* Individuals who had not to get vaccinated
* Individuals whose physical activity level is between 600-3000 MET min/week according to the IPAQ-SF (sedentary)

Exclusion Criteria:

* Individuals who are hospitalized and treated for COVID-19
* Individuals with previously diagnosed Chronic Obstructive Pulmonary Disease (COPD), heart disease, and/or rheumatic diseases
* Individuals who have had surgery in the last six months

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Quadriceps femoris strength | Once time, 3 minutes
  To measure the knee extension strength, the individual brings the knee from 90 degrees flexion to full extension in sitting. To standardize the test, the lower extremities will be fixed of the chair with a belt, allowing full extension of the knee. Three measurements will be performed from the distal tibia with a dynamometer, and the score will be recorded in Newtons.
Biceps brachii strength | Once time, 3 minutes
  Elbow flexion will also be measured in a sitting position in a chair. To standardize the given resistance, the upper extremity of the individual will be fixed to the arm support of the chair, allowing elbow flexion with a belt. During the measurement, the individual will try to flex the forearm in supination. Meanwhile, three measurements will be taken from the distal forearm with a dynamometer. The average score will be recorded in Newtons.
Upper extremity flexibility-Back scratch test | Once time, 3 minutes
  The back-scratch test evaluates upper extremity flexibility. The individual will externally rotate one arm over her/his shoulder to reach the lowest point on the back with the palm facing the back. The other extremity reaches the highest point on the back with the palm facing forward by internal rotation of the other arm. The distance between the middle fingers of both hands will be measured with a tape measure. If the middle fingers do not touch each other, the distance between them is recorded as a minus value in centimeters, if fingers can reach completely, as a zero value, if the fingers cross each other, as a positive value in centimeters
Lower extremity flexibility-Sit and reach test | Once time, 2 minutes
  Sit and reach test evaluates lower extremity flexibility. In the test, a sit and reach board with 30 cm height, 45 cm width, and 100 cm length is used. The "0" reference point is taken as the 25 cm inner part where the feet are placed on the sit and reach the board. The part closer to the individual from the reference point shows negative values, and the part towards the far side shows positive values. Individuals will reach as far as with their fingertips by placing their feet on a sit-and-reach board. The test is repeated three times. The average score is recorded
Functional strength of trunk muscles-Sit-ups test | Once time, 2 minutes
  The sit-ups test is a measure the endurance of the abdominal and hip-flexor muscles. The physiotherapist will fix the feet and ask the individuals to do trunk flexion in the knee flexion position. The number of movements performed for 30 seconds will be recorded.
Functional strength of trunk muscles-Push-ups test | Once time, 2 minutes
  The test will be in the prone position, with the hands at shoulder level and the elbows flexed, positioned near to the body. Individuals will raise the head, shoulders, and trunk from the ground with their elbows in full extension. The test is performed with the knees in full extension for men and modified knees in flexion for women. The number of movements performed for 30 seconds will be recorded.
Muscle Endurance-Lateral bridge test | Once time, 5 minutes
  Lateral bridge test involves static, isometric contractions of the lateral muscles on each side of the trunk that stabilizes the spine. Higher scores indicate a good level of endurance.
Muscle Endurance- Biering-Sorensen test | Once time, 5 minutes
  The test measuring how many seconds the individual can keep the unsupported upper body (from the upper border of the iliac crest) horizontal, while placed prone with the buttocks and legs fixed to the couch by three wide canvas straps and the arms folded across the chest. Higher scores indicate a good level of endurance.
Muscle Endurance-Trunk flexors endurance test | Once time, 5 minutes
  Trunk flexion test involving a static, isometric contraction of the anterior muscles, stabilizing the spine until the individual exhibits fatigue. The researcher stops the test when the individual cannot hold the assumed position. Higher scores indicate a good level of endurance.
Muscle Endurance- Prone bridge test | Once time, 5 minutes
  The prone bridge test measures the muscular endurance of the abdominal muscles. Higher scores indicate a good level of endurance.
Static balance | Once time, 5 minutes
  Single leg stance test Individuals bend one knee and place the sole on the other thigh and maintain their balance in this position. The test will be performed separately for the right and left extremities with eyes open and closed. The single-leg stance balance time was recorded as seconds.
Dynamic balance | Once time, 5 minutes
  Functional reach test The functional reach test evaluates dynamic balance and limit of stability. This test measures the distance between the length of an outstretched arm in a maximal forward reach from standing while maintaining a fixed base of support. The scoring record is centimeter. Higher scores indicate a good level of balance

SECONDARY OUTCOMES:
Fatigue-modified Borg scale | Once time, 2 minutes
  Individuals will score perceived fatigue during walking and running activities with the Modified Borg Scale. According to the scale, "0" indicates no fatigue, and a score of "10" indicates unbearable fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Yürük, Assoc.Prof, Principal Investigator — Baskent University
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No